CLINICAL TRIAL: NCT04287296
Title: Providing Mental Health Support Through an Educational and Entertaining Breakfast Show in the United Kingdom - a 12-week Feasibility Trial of Wakey
Brief Title: A 12-week Feasibility Trial of a Mental Health Breakfast Show Wakey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Method X Studios Ltd (Industry)
Collaborators: Guy's and St. Thomas' Charity (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Wakey
Record Dates: First submitted 2020-02-21; First posted 2020-02-27 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Mental Wellbeing
Keywords: mental health; mental wellbeing; wellbeing; edutainment; brekfast show; feasibility study
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A non-randomised feasibility trial with all participants receiving the intervention (the breakfast show) via app that is available for free to download on iOS and Android operating systems.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App users (Experimental): The app users who are at least 18 years old.
  Interventions: Behavioral: Wakey!

INTERVENTIONS:
Behavioral: Wakey! — Everyone who has downloaded the app will receive a 9-minute morning show as an alternative to an alarm clock every Mon-Fri for 12 weeks. The show is presented by a cast of presenters who appeal to the target demographic. The intervention content is theory and evidence led, drawing on approaches from cognitive and third-wave psychotherapies, positive psychology interventions (such as those based on resilience training and growth mindset), and lifestyle mental health interventions. Additional content will be provided on the app to support the theory and techniques that are covered in the show. Fun content will also be posted in an ad-hoc manner that complement the shows or relate to cultural dates and aim to increase engagement. Wakey! will avoid any polarising topics such as politics, religion and folk science. There are several features beside the show itself: a moderated live chat between 6-9AM, feedback for users (e.g. how many days they have seen the show, current energy levels).

SUMMARY:
The aim of Wakey! is to increase access to wellbeing support to lower socio-economic groups who have traditionally been excluded from the design and evaluation of digital mental health interventions. This feasibility study is designed to explore engagement, initial efficacy and experience of using Wakey! in the underserved populations in the United Kingdom. This will be used to further adapt and refine the intervention, so it is appealing and effective in the target populations.

DETAILED DESCRIPTION:
Mental health conditions are a considerable burden for patients and health services and have been shown to have social patterning in severity and incidence. Children and adults living in the lowest 20% income bracket are two to three times more likely to develop a mental health condition than those people living in the top 20% bracket. Unemployment, working in jobs with low pay and insecure work have been found to be detrimental to mental health. Mental health services are struggling to cope with demands on services, and unequal access to support is further exacerbating health inequalities.

Digital interventions have been proposed as a solution to address the high demand for mental health support in the context of the crisis in healthcare services. These interventions provide the potential to reduce health disparities, by providing personalised low-cost infinitely reusable resource that can increase access to health interventions. However, these interventions may increase inequity, where access and usability for disadvantaged groups remain barriers. To ensure health inequalities are not further exacerbated, there is a need to develop digital interventions that are appealing and accessible those from lower socioeconomic groups. These are social groups that currently look to entertainment to regulate difficult emotions and for education.

An initial pilot of the 9-minute show was trialled in the United Kingdom with a lower socio-economic group and was well received. The app was advertised through the companies that partner with Lost In TV Audience Services, who has a database of 450,000 people. In the initial pilot 43,000 people opened the email about the app. The live morning breakfast show that ran for two weeks was used by 450 participants. The findings were that 50% watched all 10 shows, 65% said that would download the app "today", 70% said it was easier to get out of bed, 53% saw an increase in life satisfaction, and 67% reported an increase in self-efficacy.

The primary objectives of the feasibility study are:

* To assess how many people download the app in the target population
* To assess participant's engagement with the app over the 12-week trial period

The secondary objectives are:

* To explore efficacy data on Office for National Statistics well-being outcomes, sleep and self-efficacy outcomes and to see if there are any changes throughout the trial
* To explore, quantitatively and qualitatively, participants' experiences of using Wakey!

ELIGIBILITY:
Inclusion Criteria:

* App users who are at least 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3993 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-05-21 (Actual)

PRIMARY OUTCOMES:
Overall engagement | 12 weeks; collected daily (not on weekends) throughout the trial
  Number of episodes (livestream/archived) watched over the 12-week period.

SECONDARY OUTCOMES:
Change in personal well-being | 12 weeks; baseline, then weekly follow-ups until the end of the trial
  UK's national personal well-being measures (used in the Annual Population Survey) about life satisfaction, feeling the things done in life are worthwhile, happiness and anxiety. The participants are asked to rate the four domains on a scale of 0 ("not at all") to 10 ("completely"). Higher scores indicate higher perception of wellbeing (except for anxiety, where higher scores indicate higher level of anxiety).
Change in the ease of getting up in the morning | 12 weeks; baseline, then weekly follow-ups until the end of the trial; as a daily question from Mon-Fri during the trial
  The participants are asked to rate how easy it was to get up this morning on a scale of 0 ("not at all") to 10 ("completely").
Change in self-efficacy | 12 weeks; baseline, then weekly follow-ups until the end of the trial
  The participants are asked to assess to what extent they agree with the statement "I can successfully overcome life's daily challenges". The answers include: strongly agree (1), agree (2), neither agree or disagree (3), disagree (4), strongly disagree (5). Higher scores indicate lower self-efficacy.
Entertainment value of the episode | 12 weeks; daily question from Mon-Fri during the trial
  The participants are asked to rate how entertaining did they find the current episode on a scale of 0 ("not at all") to 10 ("completely").

CONTACTS AND LOCATIONS:
Locations (1):
- Method X Studios, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oeren M, Jordan I, Coughlin D, Turnbull S. Improving Access to Behavioral Strategies to Improve Mental Well-being With an Entertaining Breakfast Show App: Feasibility Evaluation Study. JMIR Form Res. 2022 Mar 23;6(3):e25715. doi: 10.2196/25715. PMID 35319468